CLINICAL TRIAL: NCT06651944
Title: Invisalign® System with Mandibular Advancement Featuring Occlusal Blocks (MAOB) Post-Market Study
Brief Title: Invisalign® System with Mandibular Advancement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A005541
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Class II Malocclusion; Mandibular Advancement; Mandibular Retrognathism; Excessive Overjet
Keywords: Class II Malocclusion; Mandibular Advancement; Invisalign; Orthodontics; Occlusal Blocks; Growing Patients
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Invisalign® System with Mandibular Advancement (Experimental): all participants will receive the study device
  Interventions: Device: Invisalign® System with mandibular advancement featuring occlusal blocks

INTERVENTIONS:
Device: Invisalign® System with mandibular advancement featuring occlusal blocks — Class II correction using the Invisalign® System with mandibular advancement featuring occlusal blocks

SUMMARY:
The goal of this clinical trial is to observe study participants' comfort and fit of their aligners with occlusal blocks, as well as evaluate the engagement of the blocks using the Invisalign® System with mandibular advancement featuring occlusal blocks

ELIGIBILITY:
Inclusion Criteria:

• Subject must be eligible for Invisalign treatment with mandibular advancement

Exclusion Criteria:

* Subject's dentition not compatible with device or allergy to device materials
* Subject who is pregnant, has active caries, periodontal disease, TMD, root resorption, has HAE (hereditary angioedema), has been diagnosed with epilepsy or any other seizure disorder

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comfort and fit | Through the study completion of up to 2 years
  Measured using quality of life surveys at the insertion, interim, and end of study visits. Measured on a scale which the subject rates from 1-Always to 5-Never on their current experience.

SECONDARY OUTCOMES:
Class II correction | Through the study completion of up to 2 years
  measured through analysis of intraoral scans

OTHER OUTCOMES:
Class II correction | Through the study completion of up to 2 years
  measured through analysis of cephalometric radiographs

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Astra Orthodontics, Richmond, British Columbia
  - MacKenzie Orthodontics, Saint John, New Brunswick
  - Discover Orthodontics, Brampton, Ontario

IPD SHARING:
Plan to Share IPD: No
Data is planned to be shared with Sponsor and Investigators only